CLINICAL TRIAL: NCT01420575
Title: Using a Visual Decision Aid (DA) to Facilitate Shared Decision Making (SDM) During Antipsychotic Treatment in Schizophrenia.
Brief Title: Decision Aid to Facilitate Shared Decision Making During Treatment in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment rate.
Sponsor: VA Nebraska Western Iowa Health Care System (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Nebraska Educational Biomedical Research Association (Unknown)
Responsible Party: Principal Investigator, SRIRAM RAMASWAMY, Staff Psychiatrist, VA Nebraska Western Iowa Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAM-00730
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Shared Decision; Decision Aid; Antipsychotic; Weight Gain; Olanzapine; Lexapro; Perphenazine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Weight Gain | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visual Decision Making Aid (Experimental): Shared decision-making, in contrast to traditional medical decision-making, involves a collaborative process where patients discuss personal values and preferences and clinicians provide information to arrive at an agreed upon treatment decision. The focus of the intervention is to empower overweight patients with schizophrenia/schizoaffective disorder and help them efficiently arrive at a treatment decision that can be successfully implemented.
  Interventions: Behavioral: Visual Decision Aid and Shared Decision Making Model
- Usual Care (Active Comparator): Usual care reflects the standard of care in psychiatry. Psychiatrists will recommend treatment for overweight patients with schizophrenia on olanzapine who have failed to lose weight despite life style and dietary modifications. They may recommend switching to a comparable antipsychotic with a lower incidence of weight gain.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Visual Decision Aid and Shared Decision Making Model — Visual aid is a graph showing the average weight of patients who take olanzapine versus perphenazine over the course of 18 months. A script explaining the information on the graph, accompanies the graph. Patient may decide to stay on current dose of olanzapine, or be tapered off and prescribed a dose of perphenazine based on current symptoms and tolerability. Perphenazine (4-8mg ORALLY 3 times a day) will be used.
  Other Names: Zyprexa
  Arms: Visual Decision Making Aid
Behavioral: Usual Care — Usual care is standard clinical discussion and advice from a psychiatrist. Patient may decide to stay on current dose of olanzapine, or be tapered off and prescribed a dose of perphenazine based on current symptoms and tolerability. Perphenazine (4-8mg ORALLY 3 times a day) will be used.
  Other Names: Zyprexa
  Arms: Usual Care

SUMMARY:
We hypothesize that the use of a visual decision aid tool to educate patients regarding potential harm with respect to weight gain with olanzapine versus perphenazine can lead to better shared decision making by patients, increase rates of antipsychotic switches and promote weight loss in overweight patients with schizophrenia/schizoaffective disorder.

Our specific aims are the following:

1. To investigate the effects of a visual decision aid, versus care as usual, on patients' perceived difficulties in medical decision making regarding switching antipsychotics in overweight veterans with schizophrenia or schizoaffective disorder.
2. To investigate the effects of a visual decision aid and a shared decision making model on rate of medication switches (from olanzapine to perphenazine) in overweight veterans with schizophrenia or schizoaffective disorder.
3. To investigate the effects of a visual decision making aid and shared decision making model on BMI in overweight veterans who switch from olanzapine to perphenazine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of Schizophrenia or Schizoaffective Disorder as per by their medical record diagnosis.
* Patients currently on olanzapine therapy and BMI >29.9.
* Patients treated with olanzapine for greater than or equal to 3 months prior to enrollment.
* Patient would be required to have either attempted dietary, lifestyles modifications and/or participated in weight loss programs.
* Patients with no history of psychiatric hospitalizations in past six months and judged by treating clinician to be suitable for antipsychotic medication switch.
* Patients with adequate decisional capacity to make a choice about participating in this research study.
* Patients, who are able to comprehend and satisfactorily comply with protocol requirements and have an ability to read and write English.
* Patients, who signed the written consent given prior to entering any study procedure.

Exclusion Criteria:

* Patients with a history of treatment resistant schizophrenia or past trials with clozapine.
* Patients with a concurrent DSM-IV diagnosis of PTSD as per their medical record.
* Substance Dependence or Abuse (excluding nicotine) within one month prior to the screening visit.
* Patients with a history of non-response, intolerance or hypersensitivity ot perphenazine.
* Subjects with history of treatment of clozapine.
* Patients who based on history of mental status examination have a significant risk of committing suicide.
* Patients who are homicidal or violent and who are in the Investigator's opinion in significant imminent risk of hurting others.
* Female patients who are pregnant, planning to become pregnant, or if of childbearing potential, not using an acceptable method of birth control.
* Patient currently receiving depot neuroleptics.
* Patients with visual impairments.

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Differences in Decisional Conflict scores between the two groups (intervention versus care as usual) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Ramaswamy, M.D., Principal Investigator — Department of Veterans Affairs/NWIHCS; Robert Rosenheck, M.D., Principal Investigator — Department of Veterans Affairs/NWIHCS
Locations (1):
- Omaha Veterans Affairs Medical Center, Omaha, Nebraska, United States